CLINICAL TRIAL: NCT06130878
Title: Effects of a Rhythmic Exercise Program on the Physical, Mental and Cognitive Performance of Older Adults With Cognitive Impairment.
Brief Title: Rhythmic Exercise in Older Adults With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: -UJAEN
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (No Intervention): This group does not receive any treatment.
- EXPERIMENTAL GROUP (EG) (Experimental): People assigned to this group will undergo a 12-week physical training intervention
  Interventions: Other: Rhythmic exercise

INTERVENTIONS:
Other: Rhythmic exercise — A multicomponent rhythmic physical training will be carried out, with a predominance of QMT, following the principles of "Animal Flow" [46] and including the following components: wrist mobilizations; activations; specific stretching positions; special locomotor movements or "traveling forms"; interruptions and transitions with dynamic movements and choreographic sequences of "Flow". Aspects related to the control of intensity, volume and progression strategy have yet to be defined.
  Arms: EXPERIMENTAL GROUP (EG)

SUMMARY:
Rhythmic physical exercise is a very promising non-pharmaceutical tool to prevent or reduce cognitive decline that occurs in people sixty years of age or older. The main objective is to determine the effect of a rhythmic exercise program on the physical, mental and cognitive performance of older adults with cognitive impairment. The main variables of the study will be: global cognitive function evaluated by the Mini Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MoCA); attention and executive functions evaluated using the Trail Making Test (TMT) part A and B. As secondary variables, the functional abilities evaluated using the Senior Fitness Test (SFT) will be taken into account. Additionally, sociodemographic variables and variables related to health status will be evaluated. These will take into account the quality of sleep evaluated with the Pittsburgh index, the nutritional status evaluated using the Mini Nutritional Assessment-Short Form (MNA-SF) scale, and the Stress and anxiety levels will be assessed using the Depression Anxiety Stress Scales-21 (DASS-21). All variables will be evaluated before the intervention and after it. After the intervention, it is expected that the exercise program will improve the neurocognitive performance, as well as the functional and psychological abilities of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years old or older
* Do not participate in any physical exercise program
* Present physical autonomy to participate in the physical activities required by the study.
* Present scores of > 25 on the MMSE
* Present current affiliation to the social health security system.
* Sign the informed consent
* Understand the instructions, programs and protocols of this project.
* Complete more than 90% of the intervention with exercise.

Exclusion Criteria:

* Present medical contraindications for performing physical tests.
* Present diseases that limit cognitive performance and physical activity.
* Present vestibular diseases
* Present rheumatological diseases that can be exacerbated by stress articulate.
* Refusing to sign the informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
MoCA (Montreal Cognitive Assessment) | Up to twelve weeks
  Instrument that examines the skills of attention, concentration, executive functions, memory, language, visuoconstructive abilities, calculation and orientation and the maximum score is 30.
TMT (Trail Making Test) | Up to twelve weeks
  It is used to assess executive function. It measures timed motor and visual tasks, and is divided into two tests: Part A (TMTA), which assesses speed and psychomotor attention and requires connecting consecutively numbered circles; and Part B (TMTB), which tests executive function and requires connecting alternating circles of numbers and letters. Longer completion times indicate poor performance.
Mini-Mental State Examination (MMSE) | Up to twelve weeks
  The most widely used cognitive screening test to assess suspected symptoms consistent with cognitive impairment or dementia. Written test with a maximum score of 30. The cut-off point established for the MMSE defines "normal" cognitive function is generally set at 24, lower scores indicate more serious cognitive problems.
SFT (Senior Fitness Test) | Up to twelve weeks
  Instrument used to assess functional abilities. It consists of the following tests: muscle strength (upper and lower limbs), aerobic endurance, flexibility (upper and lower limbs) and agility, 6-minute walk test, Sit-to-foot test using a chair (measures flexibility of the lower body, Try to clasp hands behind your back, Try to get up, walk 8 feet and sit back.
The Short Form-36 Health Survey (SF-36) | Up to twelve weeks
  Used extensively for assessing health-related quality of life. The results are values between 0 and 100. Optimal health is represented by scores of 100 and very poor health would equal 0.
Chair sit and reach test | Up to twelve weeks
  To test low back and hamstring flexibility.
Back scratch test | Up to twelve weeks
  To measure general shoulder range of motion.
PSQI (Pittsburgh Sleep Quality Index) | Up to twelve weeks
  A simple and valid assessment of both sleep quality and disturbance that might affect. They consist of 10 questions divided into four subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep discomfort, medication use and daytime dysfunctions, adding up to a total score. The higher value represents a worse result. Higher scores indicate poorer sleep.
The Yesavage Geriatric Depression Scale | Up to twelve weeks
  Questionnaire used to screen for depression in older people. Scores from 00 to 05 indicate Normal screening, 06 to 10 Moderate Depression screening, and 11 to 15 Severe Depression screening.

SECONDARY OUTCOMES:
Tinetti scale | Up to twelve weeks
  It is used to determine early the risk of falling in an elderly person during the year following its application. The result of both sections will be added, so that a score of less than 19 points will imply a high risk of falls, a score of 19 to 24 will reflect medium risk of falls and a score of 25 to 28 will indicate low risk of falls.
Frailty phenotype | Up to twelve weeks
  Five original characteristics are evaluated: involuntary weight loss, self-reported exhaustion, slow gait speed, weakness, and low physical activity.
Handgrip Strength | Up to twelve weeks
  Dynamometer will be employed to assess hand grip strength.
Mindful Attention Awareness Scale (MAAS) | Up to twelve weeks
  It evaluates, in a global way, the dispositional capacity of an individual to be attentive and aware of the experience of the present moment in everyday life. The scale is a 15-item univariate self-report with a view of the mindfulness construct centered on the attention / consciousness variable.

CONTACTS AND LOCATIONS:
Locations (1):
- U.E.D. Virgen de la Capilla, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No